CLINICAL TRIAL: NCT01189019
Title: High Dose Lucentis for Persistent Pigment Epithelial Detachment in Neovascular Age-related Macular Degeneration - The HiPED Study
Brief Title: HiPED - High Dose Lucentis for Persistent Pigment Epithelial Detachments in Age-related Macular Degeneration
Acronym: HiPED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug dose became unavailable
Sponsor: Anne Fung MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Anne Fung MD, Principal Investigator, Pacific Eye Associates
Organization: Pacific Eye Associates (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4928
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Wet Macular Degeneration; Macular Degeneration; Retinal Pigment Epithelial Detachment
Keywords: ranibizumab; Wet macular degeneration; macular degeneration; PED; Retinal Pigment Epithelial Detachment
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Retinal Detachment | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - 2mg ranibizumab monthly (Experimental): 2mg ranibizumab monthly
  Interventions: Drug: ranibizumab
- Group 2 - 2mg x 3 then PRN (Active Comparator)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 2mg intravitreal injection monthly
  Arms: Group 1 - 2mg ranibizumab monthly
Drug: ranibizumab — 2mg monthly x 3 doses, then as needed based on recurrence of activity on OCT
  Arms: Group 2 - 2mg x 3 then PRN

SUMMARY:
In this fifth year of anti-VEGF therapy for neovascular AMD, retinal physicians are collecting groups of patients who either do not or only partially respond to anti-VEGF therapy. This study will evaluate the efficacy and safety of 2mg ranibizumab specifically for patients with fibrovascular PEDs that have not resolved following at least 6 consecutive injections of ranibizumab or bevacizumab over the previous 12 months. The investigators hypothesize that the 2mg dose will be able to completely eliminate the persistent PEDS in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Active or recurrent neovascular age-related macular degeneration involving the fovea on FA
* Presence of persistent fibrovascular pigment epithelial detachment on OCT following a minimum 6 previous treatments in previous 12 months with ranibizumab and/or bevacizumab. Patients may have received more than 12 months of anti-VEGF therapy.
* ETDRS Best Corrected Visual acuity 20/32 - 20/400

Exclusion Criteria:

* Prior treatment with verteporfin, or external-beam radiation therapy, or transpupillary thermotherapy, Previous subfoveal focal laser photocoagulation involving the foveal center, History of vitrectomy, submacular surgery, or other surgical intervention for AMD, Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals) in study eye.
* Lesion Characteristics: Subfoveal fibrosis or atrophy in study eye, CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia.
* Concurrent Ocular Conditions: Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma), Any concurrent intraocular condition in the study eye (e.g., diabetic retinopathy or glaucoma) that, in the opinion of the investigator, could either, Require medical or surgical intervention during the 12-month study period to prevent or treat visual loss that might result from that condition, or If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 12-month study period, Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure 30 mmHg despite treatment with anti-glaucoma medication)

Concurrent Systemic Conditions

* Pregnancy or premenopausal women not using adequate contraception The following are considered effective means of contraception: surgical sterilization; use of oral contraceptives; barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel; an IUD; or contraceptive hormone implant or patch.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications

Other

* Inability to dilate pupils sufficient for adequate fluorescein angiography
* Inability to comply with study or follow up procedures

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test)
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mean change in visual acuity from baseline to 24 months | 24 months
  Best corrected visual acuity on the ETDRS chart at 4 meters will be compared

SECONDARY OUTCOMES:
Visual acuity from baseline to 6 months | 6 months
  BCVA on ETDRS will be compared from baseline to 6 months
Safety | 12 months
  incidence and severity of ocular and non-ocular adverse events will be evaluated through 12 months
% with > 15 ETDRS letter gain from baseline through 12 months | 12 months
Change in OCT CST from baseline through 6 and 12 months | 12 months
Time to recurrence of PED in PRN Arm | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fung, MD, Principal Investigator — Pacific Eye Associates / California Pacific Medical Center
Locations (3):
- United States (3):
  - Pacific Eye Associates, San Francisco, California
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Tennessee Retina, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Presented at medical conferences, manuscript in preparation

REFERENCES:
- See also: Pacific Eye Associates — http://www.pacificeye.com
- See also: Retina Associates of Kentucky — http://www.retinaky.com/